CLINICAL TRIAL: NCT05200052
Title: Effect of Colchicine Use On Left Ventricle Systolic Function Using Speckle Tracking Echocardiography in Patients With Anterior S-T Segment Elevation Myocardial Infarction
Brief Title: Effect of Colchicine On Left Ventricle Function After Anterior Myocardial Infarction Assessed By Speckle Tracking
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Mohamed Radwan, Principal investigator, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FMASUMD88/2020
Record Dates: First submitted 2021-12-20; First posted 2022-01-20 (Actual); Last update posted 2022-08-23 (Actual); Status verified 2022-08

CONDITIONS: Anterior MI; Colchicine
MeSH Terms: conditions — Anterior Wall Myocardial Infarction | interventions — Colchicine; Tablets

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Colchicine 0.5 mg oral tablet (Active Comparator): 100 patients presented with anterior Myocardial infarction undergoing primary Percutaneous coronary intervention will receive colchicine tablet 1mg loading dose and colchicine 0.5 mg maintance dose for 6 months and will do longitudinal strain pattern echocardiography to asses left ventricles systolic function
  Interventions: Drug: Colchicine 0.5 mg Oral Tablet
- Standard anti ischemic treatment (No Intervention): 100 patients presented with anterior myocardial infarction undergoing primary percutaneous coronary intervention will do longitudinal strain pattern echocardiography to asses left ventricles systolic function

INTERVENTIONS:
Drug: Colchicine 0.5 mg Oral Tablet — Colchicine loading dose 1 mg and maintenance dose 0.5 mg for 6 months in addition to standard anti ischemic treatment.
  Other Names: Standard anti ischemic treatment
  Arms: Colchicine 0.5 mg oral tablet

SUMMARY:
Effect of colchicine use on Left ventricles systolic function in patients with anterior S-T elevation myocardial infarction undergoing primary Percutaneous coronary intervention by using speckle tracking Echocardiography longitudinal strain pattern

DETAILED DESCRIPTION:
The study participants are patients presented with anterior myocardial infarction.

They will be divided into 2 groups. The first group will receive colchicine loading dose of 1mg then 0.5 mg maintenance dose in addition to the standard anti ischemic treatment for 6 months.

The other group will only receive the standard anti ischmic treatment. Speckle tracking echocardiography will be done to all patients to assess left ventricular longitudinal strain pattern.

ELIGIBILITY:
Inclusion Criteria:

▪︎Anterior S-T segment elevation myocardial infarction with time of presentation less than 12 hours.

Exclusion Criteria:

* Severe renal impairment.
* Cardiac arrest.
* Cardiogenic shock.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2022-08-01 (Actual); Study Completion 2022-08-01 (Actual)

PRIMARY OUTCOMES:
Average of global longitudinal strain pattern | 6 months
  Assessment of left ventricular longitudinal strain by speckle tracking echocardiography after beforr and after colchicine

SECONDARY OUTCOMES:
Number of mortality during study | 6 months
  Death from any cause

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Radwan, Master, Principal Investigator — Ain Shams University
Locations (1):
- Ain Shams University hospitals, Cairo, Egypt